CLINICAL TRIAL: NCT05853796
Title: Observational Dutch Young Symptomatic StrokE studY - Extended
Brief Title: Observational Dutch Young Symptomatic StrokE studY - nEXT
Acronym: ODYSSEY-nEXT
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Synapse bv (Industry)
Responsible Party: Sponsor
Other Study IDs: NL77518.091.21
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Ischemic Stroke; Stroke in the Young; Cardiovascular Diseases; Cerebrovascular Disorders; Embolism and Thrombosis; Thrombophilia; Coagulation
MeSH Terms: conditions — Ischemic Stroke; Cardiovascular Diseases; Cerebrovascular Disorders; Embolism and Thrombosis; Thrombophilia; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients and controls at baseline:
  1 x 2.7 mL + 1 x 9ml sodium citrate tube, aliquoted in 4 x 1000 µL cryovials;
  1 x 5 mL serum tube, aliquoted in 3 x 500 µL sterile cryovials;
  1 x 3 mL EDTA tube, aliquoted in 3 x 500 µL cryovials;
  For 20 patients and 20 controls from the Radboudumc the following tubes were addionally collected for whole blood analysis:
  1x 2.7 ml citrate tube 3 x 10 ml EDTA tube for PBMCs isolation and storage.
  Patients at 3-month visit:
  1 x 2.7 mL + 1 x 9ml sodium citrate tube, aliquoted in 4 x 1000 µL cryovials;
  1 x 5 mL serum tube, aliquoted in 3 x 500 µL sterile cryovials;
  1 x 3 mL EDTA tube, aliquoted in 3 x 500 µL cryovials;
  For 20 patients and 20 controls from the Radboudumc the following tubes were addionally collected for whole blood analysis:
  1x 2.7 ml citrate tube 3 x 10 ml EDTA tube for PBMCs isolation and storage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with acute ischemic stroke at young age (18-50 years): Patients aged 18 to 50 years with first-ever ischemic stroke or transient ischemic attack.
- Healthy controls: Healthy controls (aged 18 to 50 years) without cardiovascular diseases in their medical history. Subjects age- and gender-matched to patients

SUMMARY:
BACKGROUND: Worldwide, 2 million patients aged 18-50 years suffer an ischemic stroke each year with an increasing trend over the past decade due to yet unknown reasons. Whereas prognosis and antithrombotic treatment in older patients with cardiovascular disease are among the best studied topics in clinical medicine, this does not hold true for patients at young age. It is of great importance to treat these patient groups correctly to prevent recurrence and bleeding complications. However, previous research have shown that there is a long-term increased risk of recurrent ischemic events despite the secondary prevention and a subsequent increased bleeding risk. To tailor effective antithrombotic therapy to the individual patient, it is essential to understand the underlying pathogenesis and identify modifiable risk factors in young patients for recurrence or bleeding. It is thought that abnormalities of hemostasis may play a key role in early-onset ischemic stroke. First, prothrombotic conditions are associated with an increased risk for ischemic stroke at young age. In addition, disturbance of the hemostatic balance due to one or several triggers can activate the coagulation cascade, which on its turn can lead or contribute to clot formation and subsequent arterial occlusion. In previous study, there were indications that trigger factors such as fever and/or an infection in the days prior to the stroke may play a role in the pathogenesis. This suggests that an interaction between inflammation, endothelial damage and coagulation may lead to the formation of a clot. In this observational study we aim to investigate the role of the immune system, endothelial damage and coagulation in the pathogenesis and prognosis of stroke in young patients.

OBJECTIVE: To investigate the role of hemostasis, inflammation and endothelial activation in the etiology and prognosis in an acute ischemic stroke (or TIA) in young stroke patients.

STUDY DESIGN: Multicentre prospective observational study

STUDY POPULATION:

All patients aged between 18 and 50 years old with a first-ever ischemic stroke or TIA who are admitted to the neurology ward or seen at the outpatient clinic of one of the participating centers.

Main exclusion criteria are: history of clinical TIA, ischemic stroke or intracerebral hemorrhage. A intracerebral hemorrhage resulting from trauma, known aneurysm or underlying intracerebral malignancy. A venous infarction, retinal infarction and amourosis fugax. Inadequate control of the Dutch language to reliably sign an informed consent from and/or participate in the follow-up. Patients are excluded if they have a contra indication for 3T MRI.

In addition 60 healthy controls (18-50 years old) will be included.

MAIN STUDY ENDPOINTS:

1. Baseline and 3 months coagulation profile:

   Whole blood and platelet poor plasma thrombin generation, platelet function tests, and coagulation biomarkers, screening for thrombophilia.
2. Baseline and 3 months inflammation/endothelial activation profile:

   Cytokines/chemokines, expression of receptors/cofactors related to hemostasis on peripheral blood mononuclear cells (PBMCs), stimulation tests of PBMC's to assess trained immunity.
3. Vessel wall enhancement on 3 Tesla MRI
4. Questionnaire trigger factors

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first-ever transient ischemic attack (TIA) or acute ischemic stroke aged between 18 and 50 years old
* For this study, acute stroke is defined as "occurence of acute neurological deficit lasting more than 24 hours, with confirmation on imaging (CT(-a) or MR(-a))".TIA is defined as "occurence of acute neurological deficit lasting less than 24 hours with confirmation of ischemia on MRI).
* Patients have a kidney function eGFR>30ml/min.

Exclusion Criteria:

* A history of clinical TIA, ischemic stroke or intracerebral hemorrhage
* A intracerebral hemorrhage resulting from trauma, known aneurysm or underlying intracerebral malignancy.
* A venous infarction, retinal infarction or amourosis fugax.
* Inadequate control of the Dutch language to reliably sign an informed consent from and/or participate in the follow-up
* Patients are excluded if they have a contra indication for 3T MRI.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patients aged 18 to 49 hospitalized due to first-ever imaging-positive ischemic stroke or transient ischemic attack.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2037-01-01 (Estimated)

PRIMARY OUTCOMES:
Difference of concentration biomarkers and coagulation assays between patients and controls | At baseline and 3 month visit
  Biomarkers and assays of coagulation, inflammation and endothelium activation

SECONDARY OUTCOMES:
Nonfatal or fatal recurrent cardiovascular (ischemic) events | 10 years
  Ischemic stroke or transient ischemic attack, acute coronary syndrome, peripheral artery disease
Recurrent venous thrombotic events | 10 years
  Deep venous thrombosis, pulmonary embolism, cerebral venous sinus thrombosis
Death from any cause | 10 years
Malignancy | 10 years
Bleeding complications | 10 years
  Minor and major bleeding complications
Vessel wall imaging on 3T MRI | At baseline
  Detection of vessel wall enhancement on MRI in young stroke patients

OTHER OUTCOMES:
Modified Rankin Scale | at 3-month visit and at annual follow-up contacts from year 1 to year 10
  Functional outcome will be assessed with modified Rankin Scale
Functional outcome will be assessed with Barthel Index | at 3-month visit and at annual follow-up contacts from year 1 to year 10.
Coping strategies | at 3 months visit and 6 months
  Questionnaire about different strategies to cope with major setbacks.
Subjective cognitive outcome | at 6-month follow-up
  Subjective cognition will be assessed with an electronic questionnaire

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Radboudumc, Nijmegen, Gelderland
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Isala, Zwolle, Overijssel
  - HagaZiekenhuis, The Hague, South Holland
  - Medisch Centrum Leeuwarden, Leeuwarden

REFERENCES:
- [Derived] Spiegelenberg JP, Verburgt E, den Hertog H, de Laat KF, van Rooij FG, van Uden IWM, Arntz RM, van den Wijngaard IR, Kessels RPC, Piai V, van der Kolk A, Roest M, de Laat B, Middeldorp S, Tuladhar A, Leentjens J, de Leeuw FE. Role of inflammation and haemostasis on aetiology and prognosis in young patients with ischaemic stroke: study protocol of the Observational Dutch Young Symptomatic StrokE study-EXTended (ODYSSEY-nEXT) - a multicentre prospective cohort study. BMJ Open. 2025 Mar 21;15(3):e096330. doi: 10.1136/bmjopen-2024-096330. PMID 40118475